CLINICAL TRIAL: NCT01029834
Title: Treating Overweight Youth: A Family Based Approach in Primary Care
Brief Title: Treating Pre-School Children at Risk for Overweight in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Teresa Quattrin, Chief, Division of Diabetes/Endocrinology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD053773-01 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Overweight
Keywords: BMI >85%for age and gender
MeSH Terms: conditions — Overweight; Coitus | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention- Lifestyle family based (Experimental): Behavioral family based
  Interventions: Behavioral: family based lifestyle and behavioral counseling
- Information control (Active Comparator): Child intervention only
  Interventions: Behavioral: counseling focused on the child

INTERVENTIONS:
Behavioral: family based lifestyle and behavioral counseling — 16 group meetings
  Arms: Intervention- Lifestyle family based
Behavioral: counseling focused on the child — 16 meetings
  Arms: Information control

SUMMARY:
The goal of this study is to test, in the primary care setting, the efficacy of an innovative intervention program for children aged 2-5 years with a BMI over the 85th percentile and one overweight parent (BMI >27 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* 2-5 year old with a BMI greater than the 85th% for age and sex
* one overweight parent (BMI>27kg/m2)
* child with normal developmental milestones
* history of adherence to 90% of scheduled primary care visits
* parent must be at 5th grade reading and speaking of English language or the spanish language
* no plans on moving out of the area for the 2 years subsequent to enrollment

Exclusion Criteria:

* child with a height 2 SD below the mean for age and sex and/or pathological growth velocity
* SGA
* any chronic disorders influencing energy intake and/or growth
* any orthopedic disorder preventing the child or the parent from ambulation normally and performing the activity prescribed by the program
* any medication known to have the potential of affecting weight changes
* parent or child with psychiatric and/or eating disorder
* participating mother who is pregnant or planning a pregnancy
* parent being acquainted with the parent of a previously randomized study participant

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2008-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percent BMI overweight for child and parent | baseline-6,12,18, 24 months

SECONDARY OUTCOMES:
Reduction in number of sugared drinks, high energy food and sedentary activities. Increase in fruit, vegetable and physical activity | baseline, 6,12,18,24

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Quattrin, MD, Principal Investigator — University at Buffalo/Women and Children's Hospital of Buffalo
Locations (2):
- United States (2):
  - WNY urban practices, Buffalo, New York
  - WNY suburban practices, Williamsville, New York

REFERENCES:
- [Derived] Quattrin T, Roemmich JN, Paluch R, Yu J, Epstein LH, Ecker MA. Treatment outcomes of overweight children and parents in the medical home. Pediatrics. 2014 Aug;134(2):290-7. doi: 10.1542/peds.2013-4084. PMID 25049340
- [Derived] Quattrin T, Roemmich JN, Paluch R, Yu J, Epstein LH, Ecker MA. Efficacy of family-based weight control program for preschool children in primary care. Pediatrics. 2012 Oct;130(4):660-6. doi: 10.1542/peds.2012-0701. Epub 2012 Sep 17. PMID 22987879